CLINICAL TRIAL: NCT06278948
Title: Randomized Controlled Investigator Blinded Comparative Study of the Efficacy and Tolerability of Test Product Versus Cysteamine 5% in the Treatment of Facial Epidermal Melasma Over 4 Months
Brief Title: Efficacy and Tolerability of Test Product Versus Cysteamine 5% in Treatment of Facial Epidermal Melasma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cosmetique Active International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LRP23023-depigmenting cream
Record Dates: First submitted 2024-02-19; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Melasma
Keywords: facial epidermal melasma; MASI; Cysteamine 5%
MeSH Terms: conditions — Melanosis | interventions — enkephalin, Ala(2)-cysteamine(5)-

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group TP: Test Product (Experimental): Subjects (aged 20-50 years) with mild to severe facial epidermal melasma for more than 1 year
  Interventions: Other: Group TP
- Group CYS: Cysteamine 5% (Active Comparator): Subjects (aged 20-50 years) with mild to severe facial epidermal melasma for more than 1 year
  Interventions: Drug: Group CYS

INTERVENTIONS:
Other: Group TP — Application full face, twice daily, in the morning and at bedtime for 4 months
  Other Names: Test Product
  Arms: Group TP: Test Product
Drug: Group CYS — Application short contact, of thin layer once daily at bedtime for 4 months
  Other Names: Cysteamine 5%
  Arms: Group CYS: Cysteamine 5%

SUMMARY:
This interventional, randomized, investigator blinded, controlled study conducted in one centre consists in a 4-month evaluation period within the same season avoiding sunny season on 140 subjects with facial epidermal melasma.

DETAILED DESCRIPTION:
Melasma is a very common pigmentation disorder which significantly alters quality of life as per its high visibility on the face. The objective is to compare the efficacy and tolerability of the new depigmenting formulation that addresses the different targets of hyperpigmentation and includes an inhibitor of melanin production with a breakthrough innovative mechanism of action versus Cysteamine 5% in the acute management of melasma over 4 months.

Statistics:

Sample size calculation: 120 patients (60 per group) are necessary to reach the non-inferiority objective of the Test Product versus Cysteamine 5% on the modified Melasma Area and Severity Index (mMASI) change from Baseline at Month 4. To allow a rate of subjects excluded from analysis (drop out, lost to follow-up, major deviation) at Month 4, 140 subjects in total (70 per group) are enrolled.

Statistical analysis: Continuous data collected at each visit will be summarized using common statistical measures such as the count of values, mean, standard deviation, median minimum and maximum. For categorical data, summaries will be provided in terms of frequency counts (n) and percentages (%).

ELIGIBILITY:
Inclusion Criteria:

* Facial epidermal melasma (exclude mixed and dermal melasma)
* Subjects free of excessive hair, acne, cuts, abrasions, fissures, wounds, lacerations, or any other active skin conditions on the face

Exclusion Criteria:

* Subjects with any other signs of significant irritation or skin disease
* Subjects using oral contraceptive pills or hormonal implants as birth control measures during the study
* Subjects who had a skin lightening procedure in the past 8 weeks

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-10-06 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
change in mMASI scoring | from baseline to Day112
  the mMASI is calculated using 3 components: four regions of the face (forehead, right malar, left malar and chin); area of involvement for each region (using a scale from 0 to 6): darkness compared to the surrounding normal skin for each area (evaluated using a scale from 0 to 4).
change in Investigator's Global Assessment (IGA) | from baseline to Day112
  The investigator evaluates the severity of melasma using a 4-point scale (from 0 (cleared, almost cleared) to 3 (severe (markedly darker than the surrounding normal skin)).

SECONDARY OUTCOMES:
change in Subject Global Assessment of Improvement (SGAI) | from Day28 to Day112
  The subject evaluates the change on a 6-point scale from -1 (worsened) to 4 (totally cleared).

CONTACTS AND LOCATIONS:
Overall Officials: Mukta Sachdev, Principal Investigator — MS Clinical Research Pvt. Ltd
Locations (1):
- MS Clinical Research Pvt. Ltd, Bangalore, India